CLINICAL TRIAL: NCT05584748
Title: Effects of Transcranial Direct Current Stimulation (tDCS) on Cognition in Older Adults With Mild Cognitive Impairment: A Randomized Controlled Trial
Brief Title: Effects of tDCS on Cognition in MCI: A RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tung Wah College (Other)
Responsible Party: Principal Investigator, Michael Chih Chien KUO, PhD, Associate Professor, Tung Wah College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UGC/FDS17/M06/22
Record Dates: First submitted 2022-10-10; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Mild Cognitive Impairment
Keywords: tDCS; ERP/EEG; Cognition; Dorsolateral prefrontal cortex
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Simulation group (Experimental): During anodal stimulation, the participants will receive 1.5 mA of constant current over the site for 20 min, with a 15-second ramp up and scale down at the beginning and the end of the procedure.
  Interventions: Device: transcranial direct current stimulation
- Sham group (Sham Comparator): In the sham stimulation condition, the current will only be administered during the first 30 seconds and last 30 seconds of the 20-minute window.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — tDCS is planned to be administered via electrodes positioned over the left dlPFC (anodal/sham electrode) and the left supraorbital area (reference electrode).

SUMMARY:
MCI is considered an intermediate stage between normal cognitive aging and dementia. As such, improving cognitive functions of people with MCI may delay dementia onset. In recent years, tDCS, which regulates brain activity by increasing or decreasing brain tissue excitability, has become a commonly used brain stimulation method. Accumulating evidence indicates the promising effects of cognitive enhancement after tDCS over the frontal scalp regions in people with MCI (PwMCI). However, previous studies were limited by including only a self-report measure, focused on memory performance, not assessing long-term effect, and not reporting their results in follow-up. In addition, knowledge of the precise physiological consequences of tDCS on the brain tissue and related neural mechanisms in PwMCI remains rudimentary. The objectives of the proposed study, which will target PwMCI, are to investigate the effects of tDCS at the left dorsolateral prefrontal cortex on the cognitive performance and to explore the modulation of neural mechanisms associated with the use of tDCS. Forty-eight MCI participants aged over 60 years will be recruited. All participants will be assessed by Hong Kong version of Montreal Cognitive Test. Participants that meet selection criteria will be invited to the experiment. Participants will be assigned to experimental or control groups randomly. The experiment will consist of pre- and post-assessments and a 1-month follow-up assessment. Between pre- and post-assessments, participants will receive 8 sessions (2x/week for 4 weeks) of tDCS treatment (either real or sham, 20 min per session). Outcome measures include digit span test, colour trail test, verbal fluency test, Chinese version of the Verbal Learning Test , and Hong Kong version of Montreal Cognitive Assessment. Participants will also complete a computer memory task at each assessment point (performance in this task is also used as an outcome measure) and will have their brain wave recorded while completing the task. The task will require them to study and memorise Chinese characters, followed by a recognition memory test. In the study phase, participants will be required to view Chinese characters and judge whether the characters are of the animal category. In the recognition phase, participants will decide whether the characters have been seen before.

DETAILED DESCRIPTION:
Randomization and blinding Due to limited available resources and the time required to collect the data, the investigators plan to implement the experiment in 4 batches, each separated by approximately two months. Each batch will include 12 participants from the same recruiting site. Six of them will be assigned to the anodal group and the other six to the sham group, using the block randomization method provided by http://www.randomization.com. The online software generates group allocation by knowing the number of participants per block (6) and number of blocks (2). Only the principal investigator will know the group assignments. Neither the participants nor the assessors will be given the information regarding the group assignments. Each participant will be given a registration number by the Principal Investigator. The tDCS device can be set to anodal or sham status. The PI will set up the tDCS device (anodal or sham) according to the participant's registration number and group through the device's administration menu. The research associate will select the stimulation protocol by inputting the participant's registration number on the device and be blinded to the participant's group assignment when performing tDCS stimulation and other assessments.

Sample size calculation The investigators used G*Power software to estimate the number of participants required to conduct repeated measure analyses of variance (within-between interactions) using the following parameters: correlation among repeated measures = 0.5, alpha = 0.05, number of groups = 2, power = 0.9 and number of measurements = 3 (assuming the correlation between repeated measures = 0.9). Effect size f is conservatively assumed to be 0.25. Based on previous experience using tDCS on participants with dementia and previous relevant studies, the investigators assumed a retention rate of 75%. Thus, the required sample size would be 48.

Procedure This proposed investigation will use a sham-controlled, randomized controlled trial. Participants will be randomly assigned to the anodal or sham groups (in 1:1 ratio). The stimulation method (anodal/sham) will be designated as the between-subject factor (independent variable). The potential participants will be screened and those who meet the selection criteria will be invited to participate in the study. Participants will attend a baseline assessment session in which the collection of demographic information, neurocognitive assessment scores, and a computer task with EEG recorded will occur, followed by 8 sessions of anodal tDCS completed twice a week for 4 weeks. Multi-session tDCS studies usually have a varied intervention schedule from 1 to 5 sessions per week for 1 to 5 weeks. The investigators have opted for this schedule to balance the time spent on intervention with its potential effectiveness, and to encourage compliance. After the intervention, participants will receive post- and 1-month follow-up assessments which will be the same as the baseline assessment.

EEG data acquisition EEGs will be recorded from 64 Ag/AgCl electrodes (BioSemi Active Two) located on the standard scalp sites of the 10/20 system. Four electrodes will be used to monitor eye blinks and movements. Two other electrodes will be placed in the mastoids for the EEG signal to be re-referenced off-line. Scalp EEG will be recorded from F3. Curry 9 software (Neuroscan Compumedics, U.S.A), or newer, will be used for the EEG signal processing. The EEGs will be sampled at 1024 Hz, with a low-pass filter of -200 μV. Digital band-pass filtering from 0.1 Hz to 30 Hz will be applied off-line. The continuous EEG signals will be segmented into epochs, from 200 ms before the stimulus to 1500 ms after the stimulus onset, and then the baseline will be corrected to the pre-stimulus interval. The epochs with amplitude ± 75 μV will be omitted from averaging. The averaged ERPs will be computed for each participant by classifying the study epochs that are correctly identified subsequently or missed during the recognition phase. Using the Curry 9 software, these averaged ERP files will then be transformed into text files with voltage (μV) and temporal information (ms) that can be read by Microsoft Excel software. After further rearrangement and processing in Excel, the data will be transferred to SPSS software for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* inexperienced with tDCS
* normal or corrected-to-normal vision
* right-handed
* independent in activities of daily living
* no history of seizures, head injuries, migraine, epilepsy or other psychiatric or neurological conditions

Exclusion Criteria:

* taking medication or supplements known to affect cognition (such as Ginkgo)
* exhibiting symptoms of emotional disorders
* having a history of cerebrovascular surgery
* with a metal plate in their skull

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Digit span test (Wechsler & De Lemos, 1981) | 2 minutes
  Participants are presented with a random series of digits, and are asked to repeat them in the order presented.
Colour Trail Test (CTT) (D' Elia et al., 1996) | 8 minutes
  CTT1: Must be administered first and requires the respondent to connect circles in an ascending numbered sequence (1-25).
  CTT2: Must follow the CTT1 and requires the respondent to connect numbers in an ascending sequence while alternating between pink and yellow colors.
verbal fluency test (Lezak et al., 2004) | 3 minutes
  Participants produce as many words as possible from a category in 60 seconds.
Chinese version of the Verbal Learning Test (Chang et al., 2010) | 10 minutes
  Participants repeat 9 Chinese words after they are presented.
Hong Kong version of Montreal Cognitive Assessment (Yeung et al., 2014) | 15 minutes
  A screening tool for MCI
Computerized memory task | 40 minutes
  During the study phase of the memory task, the participants will view the Chinese words on a computer screen and decide whether they are from the animal category. After finishing the study/encoding phase, the participants will perform the recognition/test task. During this task, the participants will view characters and judge whether they had seen them previously in the study phase.
Event-related potential | 40 minutes
  Electroencephalograms are recorded while completing the computerized memory task

SECONDARY OUTCOMES:
Geriatric Depression Scale (Chiu et al., 1994) | 5 minutes
  This is a screening test for major depression. There are 15 items. Cut off score is 7/8.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuo MC, Liu KP, Ting KH, Chan CC. Differentiation of perceptual and semantic subsequent memory effects using an orthographic paradigm. Brain Res. 2012 Nov 27;1486:82-91. doi: 10.1016/j.brainres.2012.10.005. Epub 2012 Oct 10. PMID 23063888
- [Background] Kuo MC, Liu KP, Ting KH, Chan CC. Age-related effects on perceptual and semantic encoding in memory. Neuroscience. 2014 Mar 7;261:95-106. doi: 10.1016/j.neuroscience.2013.12.036. Epub 2013 Dec 25. PMID 24374080
- [Background] Meinzer M, Lindenberg R, Antonenko D, Flaisch T, Floel A. Anodal transcranial direct current stimulation temporarily reverses age-associated cognitive decline and functional brain activity changes. J Neurosci. 2013 Jul 24;33(30):12470-8. doi: 10.1523/JNEUROSCI.5743-12.2013. PMID 23884951
- [Background] Meinzer M, Lindenberg R, Phan MT, Ulm L, Volk C, Floel A. Transcranial direct current stimulation in mild cognitive impairment: Behavioral effects and neural mechanisms. Alzheimers Dement. 2015 Sep;11(9):1032-40. doi: 10.1016/j.jalz.2014.07.159. Epub 2014 Nov 20. PMID 25449530
- [Background] Ownby RL, Acevedo A. A pilot study of cognitive training with and without transcranial direct current stimulation to improve cognition in older persons with HIV-related cognitive impairment. Neuropsychiatr Dis Treat. 2016 Oct 25;12:2745-2754. doi: 10.2147/NDT.S120282. eCollection 2016. PMID 27822047
- [Background] Fileccia E, Di Stasi V, Poda R, Rizzo G, Stanzani-Maserati M, Oppi F, Avoni P, Capellari S, Liguori R. Effects on cognition of 20-day anodal transcranial direct current stimulation over the left dorsolateral prefrontal cortex in patients affected by mild cognitive impairment: a case-control study. Neurol Sci. 2019 Sep;40(9):1865-1872. doi: 10.1007/s10072-019-03903-6. Epub 2019 May 7. PMID 31062189
- [Background] Gomes MA, Akiba HT, Gomes JS, Trevizol AP, de Lacerda ALT, Dias AM. Transcranial direct current stimulation (tDCS) in elderly with mild cognitive impairment: A pilot study. Dement Neuropsychol. 2019 Apr-Jun;13(2):187-195. doi: 10.1590/1980-57642018dn13-020007. PMID 31285793

DOCUMENTS (2):
  • Statistical Analysis Plan (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT05584748/SAP_000.pdf
  • Informed Consent Form (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT05584748/ICF_001.pdf